CLINICAL TRIAL: NCT03886155
Title: Cardiac Amyloidosis Screening at Trigger Finger Release
Acronym: CAST
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mazen Hanna MD, Principal Investigator, The Cleveland Clinic
Other Study IDs: 18-1511
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Amyloidosis; Trigger Finger; Transthyretin Amyloidosis; Primary Amyloidosis of Light Chain Type
Keywords: Surgery; Surgical release; Biopsy
MeSH Terms: conditions — Amyloidosis; Trigger Finger Disorder; Amyloidosis, Hereditary, Transthyretin-Related; Immunoglobulin Light-chain Amyloidosis | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Trigger finger tenosynovium (may contain tenosynovial tissue and subcutaneous fat)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trigger Finger Biopsy: Biopsy of trigger finger tenosynovial tissue during trigger finger release surgery sent to pathology for amyloid-specific analysis
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — During clinically-scheduled trigger finger release surgery, soft tissue will be removed from the trigger finger tenosynovium (which may include synovial sheath and subcutaneous fat tissue) and send to pathology to be analyzed with amyloid-specific staining.

SUMMARY:
The investigators will prospectively evaluate for the presence of amyloid deposits in soft tissue samples obtained from patients undergoing trigger finger release surgery. Patients who have tissue that stains positive for amyloid will be referred to an amyloidosis specialist.

DETAILED DESCRIPTION:
A prospective study in 2001 showed that 23% (n = 47) of biopsies for idiopathic trigger finger were positive for Congo red staining but negative for ATTR and AL amyloid via immunohistochemistry. However, mass spectrometry is now the preferred method to type amyloid tissue. Trigger finger pathology involves the same flexor tenosynovium that passes through the carpal tunnel and has been biopsied to diagnose amyloidosis. Our recent study found that 10% of older patients undergoing carpal tunnel release surgery were positive for amyloidosis, with 20% of that group presenting with cardiac involvement. 60% of the amyloid-positive group had a history of trigger finger. Surgical intervention for trigger finger could provide an opportunity to screen for amyloidosis through tenosynovial biopsy.

This study will look at the prevalence of amyloidosis in patients undergoing surgical intervention for idiopathic trigger finger. The study hypothesis is at least 10% of such patients will be positive for amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years at the time of surgical biopsy.
* Undergoing surgical intervention for idiopathic trigger finger.
* Able to consent.

Exclusion Criteria:

* Known history of amyloidosis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing trigger finger release surgery
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of amyloidosis in older patients undergoing trigger finger release | Baseline to 30 days
  Incidence of amyloid deposits in soft tissue removed from trigger finger tenosynovium in older patients undergoing trigger finger release surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mazen A Hanna, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordiner-Lawrie S, Diaz J, Burge P, Athanasou NA. Localized amyloid deposition in trigger finger. J Hand Surg Br. 2001 Aug;26(4):380-3. doi: 10.1054/jhsb.2001.0571. PMID 11469845
- [Background] Sperry BW, Reyes BA, Ikram A, Donnelly JP, Phelan D, Jaber WA, Shapiro D, Evans PJ, Maschke S, Kilpatrick SE, Tan CD, Rodriguez ER, Monteiro C, Tang WHW, Kelly JW, Seitz WH Jr, Hanna M. Tenosynovial and Cardiac Amyloidosis in Patients Undergoing Carpal Tunnel Release. J Am Coll Cardiol. 2018 Oct 23;72(17):2040-2050. doi: 10.1016/j.jacc.2018.07.092. PMID 30336828